CLINICAL TRIAL: NCT03224975
Title: Acute Pain Memory Among Former Burned: Exploration of Functional Magnetic Resonance Imaging (fMRI).
Brief Title: Acute Pain Memory Among Former Burned: Exploration of fMRI.
Acronym: EXPLO-DMA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: failure to recruit
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 1708030; ID-RCB (Other: 2017-A00918-45)
Record Dates: First submitted 2017-07-13; First posted 2017-07-21 (Actual); Last update posted 2020-09-17 (Actual); Status verified 2020-04

CONDITIONS: Magnetic Resonance Imaging; Neuronal Activity
Keywords: Pain; Brain responses; Neuroimaging; fMRI; Burn; Memory
MeSH Terms: conditions — Pain; Burns

STUDY DESIGN:
Intervention Model Description: Two groups: 20 patients and 20 healthy volunteers
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- patients (Experimental): Patient who was burned will have fMRI.
  Interventions: Other: fMRI
- control group (Active Comparator): Healthy volunteers (control group) will have fMRI.
  Interventions: Other: fMRI

INTERVENTIONS:
Other: fMRI — During fMRI, patients and control group will have to thought to seven painful memories, seven emotional memories not painful, seven neutral memories. At every memory there is control test. It is to count backwards.
  Other Names: functional Magnetic Resonance Imaging (fMRI)

SUMMARY:
Pain is complex phenomenon misunderstood in spite of medical progress and neurosciences. That's why the relief of chronic pain is only partial for a lot of infection as arthrosis, chronic back pain, headaches or neuropathic pain. Certain situations bring to relive pain sensation. Investigators were interested to former burned. They wonder about somatic memory and unconscious of acute.

DETAILED DESCRIPTION:
It is a comparative and monocentric study. There are two groups. On the one hand, there is the former burned and, on the other hand, healthy volunteers. While they thought to painful memory or not, functional Magnetic Resonance Imaging (fMRI) will be performed. Then, investigators compare two functional Magnetic Resonance Imaging (fMRI).

Main objective of this study is link up between brain activity by functional Magnetic Resonance Imaging (fMRI) and acute pain memory.

ELIGIBILITY:
Inclusion Criteria:

For control group:

* Affiliated or entitled to a social security
* Have signed consent before their participation in the study
* Adult women and men french and is right handed
* Vision and hearing normal or corrected

For former burned:

* Affiliated or entitled to a social security
* Have signed consent before their participation in the study
* Adult women and men french and is right handed
* Vision and hearing normal or corrected
* Localized burn at the hand or feet onset between 12 and 24 years
* Not sequelae painful at the inclusion
* Scope and depth of the burn according to classifications CIM 10

Exclusion Criteria:

For control group:

* Any contraindications to pass an fMRI test
* Neuropathic pains and psychiatric disorders
* Medical history of head injuries
* Burn presence

For former burned:

* Any contraindications to pass an fMRI test
* Neuropathic pains and psychiatric disorders
* Medical history of head injuries

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-02-13 (Actual); Primary Completion 2019-11-25 (Actual); Study Completion 2019-11-25 (Actual)

PRIMARY OUTCOMES:
BOLD (blood-oxygen-level dependent) signal between painful memories | Months 3
  Correlation between BOLD measured by functional Magnetic Resonance Imaging (fMRI) and every conditions: painful memories, emotional memories not painful, neutral memories and control test.
BOLD (blood-oxygen-level dependent) signal between emotional memories not painful | Months 3
  Correlation between BOLD measured by functional Magnetic Resonance Imaging (fMRI) and every conditions: painful memories, emotional memories not painful, neutral memories and control test.
BOLD (blood-oxygen-level dependent) signal between neutral memories | Months 3
  Correlation between BOLD measured by functional Magnetic Resonance Imaging (fMRI) and every conditions: painful memories, emotional memories not painful, neutral memories and control test.
BOLD (blood-oxygen-level dependent) signal between control test. | Months 3
  Correlation between BOLD measured by functional Magnetic Resonance Imaging (fMRI) and every conditions: painful memories, emotional memories not painful, neutral memories and control test.

SECONDARY OUTCOMES:
BOLD (blood-oxygen-level dependent) signal between control group for every conditions | Months 3
  Correlation between BOLD measured by functional Magnetic Resonance Imaging (fMRI) and groups for every conditions: painful memories, emotional memories not painful, neutral memories and control test.
BOLD (blood-oxygen-level dependent) signal between patients for every conditions | Months 3
  Correlation between BOLD measured by functional Magnetic Resonance Imaging (fMRI) and groups for every conditions: painful memories, emotional memories not painful, neutral memories and control test.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Claude GETENET, MD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- CHU de Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No